CLINICAL TRIAL: NCT07345858
Title: Salivary Oxytocin as a Biomarker of Psychedelic Assisted Psychotherapy in Patients With Major Depressive Disorder
Brief Title: Salivary Oxytocin as a Biomarker of Psychedelic Treatment
Acronym: PAPOXT_MDD
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Tatiana Aboulafia Brakha, PhD, University of Geneva, Switzerland
Other Study IDs: BASEC ID 2025-02092
Record Dates: First submitted 2026-01-07; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: oxytocin; psychedelics; lsd; psilocybin; Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples Without DNA — Salivary samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate whether oxytocin reactivity during a psychedelic session for MDD treatment predicts treatment response, specifically by examining its relationship with changes in flexibility and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years-old
* MDD defined by DSM-V criteria, and resistant to treatment
* Ongoing classical psychotherapeutic treatment
* Agreement to discontinue necessary psychotropic medications (some classes of anti-depressants are allowed with no need to taper off).

Exclusion Criteria:

* Psychotic or bipolar disorder
* High suicidal risk
* Severe cardiovascular, hepatic or neurological (affecting the central nervous system) disorders
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be invited to participate among consecutive patients with treatment-resistant MDD enrolled for psychedelic treatment in the Division of addictology-Department of Psychiatry of the Geneva University hospitals) after receiving approval from the Swiss Federal Office of Public health for compassionate treatment with LSD or psilocybin. Only those receiving LSD or psilocybin for the first time (first treatment cycle) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Salivary Oxytocin | One day
  Measure taken during psychedelic treatment

SECONDARY OUTCOMES:
Beck Depression Inventory | 3 months
  Self-reported depressive symptoms
Cognitive Flexibility Inventory | 3 months
  Self-reported flexibility questionnaire
Trait anxiety inventory (STAI-T) | 3 months
  Self-reported anxiety symptoms
Cognitive Emotion Regulation Questionnaire (CERQ) | 3 months
  Self-reported cognitive emotion regulation strategies
Emotion Regulation Questionnaire | 3 months
  self-reported emotion regulation strategies

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided